CLINICAL TRIAL: NCT02300675
Title: Development and Evaluation of a Therapeutic Education Intervention Focused on the Accession of Patients Treated With Hormonal Therapy in the Management of Breast Cancer: PEPs Hormonotherapy
Brief Title: Therapeutic Education Intervention in Breast Cancer: PEPs Hormonotherapy
Acronym: PEPs HORMONO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-01; 2013-A00887-38 (Other: Agence Nationale de Sécurité du Médicament)
Record Dates: First submitted 2014-04-15; First posted 2014-11-25 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: therapeutic patient education; patient adherence; empowerment; breast cancer; oral adjuvant endocrine therapy; side effects
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (No Intervention): Patients follow the classic support prescription of hormonotherapy
- therapeutic education program (Experimental): Patients follow the 4 sessions of PEP hormonotherapy. The therapeutic education prgram is led by a trained educational team, inside a prevention center : Hygée centre.
  Interventions: Behavioral: therapeutic education program

INTERVENTIONS:
Behavioral: therapeutic education program
  Arms: therapeutic education program

SUMMARY:
The purpose of this study is to evaluate the feasibility and the effectiveness of a patient education program on patients' adherence to adjuvant hormone therapy (anti-estrogen or aromatase inhibitors) for breast cancer, in collaboration with teams of sociologists, patient education and medical oncologists.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* History of breast cancer
* Medical prescription for an adjuvant hormonal treatment (anti-estrogens and / or aromatase inhibitors) as monotherapy or in combination with other treatments
* Affiliated to a social security scheme

Exclusion Criteria:

* Refusal to participate, patient protected by guardianship.
* Patient unable to understand the study or unable to follow the education sessions.
* Patient with documented cognitive or psychiatric history.
* Geographical remotness (more than 100 Kms).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
measuring changes in patient compliance | 12 months
  compliance measure with prescription refillment and questionnaire. At the inclusion and at the end of the study

SECONDARY OUTCOMES:
measure of the patients' competence in the management of treatment side effects | 12 months
  measure of the patients' competence with a specific questionnaire of scenarii
Measuring the level of knowledge of patients related to the disease, the treatment and its side effects | 12 months
  Measuring the level of knowledge of patients with a specific quizz
Measuring the level of patient anxiety | 12 months
  Measuring the level of patient anxiety with HAD scale
Measuring the level of confidence of patients related to their treatment | 12 months
  Measuring the level of confidence with a visual analogic scale
patients' quality of life assessment | 12 months
  quality of life evaluated with the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Bourmaud, MD, Principal Investigator — Institut de Cancérologie de la Loire
Locations (3):
- France (3):
  - CH Lyon Sud, Pierre-Bénite
  - Hôpital Privé de la Loire, Saint-Etienne
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Golant M, Altman T, Martin C. Managing cancer side effects to improve quality of life: a cancer psychoeducation program. Cancer Nurs. 2003 Feb;26(1):37-44; quiz 45-6. doi: 10.1097/00002820-200302000-00005. PMID 12556711
- [Background] Diefenbach MA, Butz BP. A multimedia interactive education system for prostate cancer patients: development and preliminary evaluation. J Med Internet Res. 2004 Jan 21;6(1):e3. doi: 10.2196/jmir.6.1.e3. PMID 15111269
- [Background] Perol D, Toutenu P, Lefranc A, Regnier V, Chvetzoff G, Saltel P, Chauvin F. [Therapeutic education in oncology: involving patient in the management of cancer]. Bull Cancer. 2007 Mar;94(3):267-74. French. PMID 17371769
- [Background] Persijn JP, Korsten CB, Engelsman E. Oestrogen and androgen receptors in breast cancer and response to endocrine therapy. Br Med J. 1975 Nov 29;4(5995):503. doi: 10.1136/bmj.4.5995.503. No abstract available. PMID 172189
- [Background] Fisher B, Dignam J, Bryant J, DeCillis A, Wickerham DL, Wolmark N, Costantino J, Redmond C, Fisher ER, Bowman DM, Deschenes L, Dimitrov NV, Margolese RG, Robidoux A, Shibata H, Terz J, Paterson AH, Feldman MI, Farrar W, Evans J, Lickley HL. Five versus more than five years of tamoxifen therapy for breast cancer patients with negative lymph nodes and estrogen receptor-positive tumors. J Natl Cancer Inst. 1996 Nov 6;88(21):1529-42. doi: 10.1093/jnci/88.21.1529. PMID 8901851
- [Background] Rao RD, Cobleigh MA. Adjuvant endocrine therapy for breast cancer. Oncology (Williston Park). 2012 Jun;26(6):541-7, 550, 552 passim. PMID 22870539
- [Background] Lebovits AH, Strain JJ, Schleifer SJ, Tanaka JS, Bhardwaj S, Messe MR. Patient noncompliance with self-administered chemotherapy. Cancer. 1990 Jan 1;65(1):17-22. doi: 10.1002/1097-0142(19900101)65:13.0.co;2-i. PMID 2293862
- [Background] Love RR, Cameron L, Connell BL, Leventhal H. Symptoms associated with tamoxifen treatment in postmenopausal women. Arch Intern Med. 1991 Sep;151(9):1842-7. PMID 1888251
- [Background] Waterhouse DM, Calzone KA, Mele C, Brenner DE. Adherence to oral tamoxifen: a comparison of patient self-report, pill counts, and microelectronic monitoring. J Clin Oncol. 1993 Jun;11(6):1189-97. doi: 10.1200/JCO.1993.11.6.1189. PMID 8501505
- [Background] Partridge AH, Avorn J, Wang PS, Winer EP. Adherence to therapy with oral antineoplastic agents. J Natl Cancer Inst. 2002 May 1;94(9):652-61. doi: 10.1093/jnci/94.9.652. PMID 11983753
- [Background] Horwitz RI, Horwitz SM. Adherence to treatment and health outcomes. Arch Intern Med. 1993 Aug 23;153(16):1863-8. PMID 8250647
- [Background] Banning M. Adherence to adjuvant therapy in post-menopausal breast cancer patients: a review. Eur J Cancer Care (Engl). 2012 Jan;21(1):10-9. doi: 10.1111/j.1365-2354.2011.01295.x. Epub 2011 Oct 18. PMID 22004071
- [Background] Henry NL, Azzouz F, Desta Z, Li L, Nguyen AT, Lemler S, Hayden J, Tarpinian K, Yakim E, Flockhart DA, Stearns V, Hayes DF, Storniolo AM. Predictors of aromatase inhibitor discontinuation as a result of treatment-emergent symptoms in early-stage breast cancer. J Clin Oncol. 2012 Mar 20;30(9):936-42. doi: 10.1200/JCO.2011.38.0261. Epub 2012 Feb 13. PMID 22331951
- [Background] Atkins L, Fallowfield L. Intentional and non-intentional non-adherence to medication amongst breast cancer patients. Eur J Cancer. 2006 Sep;42(14):2271-6. doi: 10.1016/j.ejca.2006.03.004. Epub 2006 Apr 27. PMID 16644208
- [Background] Sant M, Allemani C, Berrino F, Coleman MP, Aareleid T, Chaplain G, Coebergh JW, Colonna M, Crosignani P, Danzon A, Federico M, Gafa L, Grosclaude P, Hedelin G, Mace-Lesech J, Garcia CM, Moller H, Paci E, Raverdy N, Tretarre B, Williams EM; European Concerted Action on Survival and Care of Cancer Patients (EUROCARE) Working Group. Breast carcinoma survival in Europe and the United States. Cancer. 2004 Feb 15;100(4):715-22. doi: 10.1002/cncr.20038. PMID 14770426
- [Result] Hohneker J, Shah-Mehta S, Brandt PS. Perspectives on adherence and persistence with oral medications for cancer treatment. J Oncol Pract. 2011 Jan;7(1):65-7. doi: 10.1200/JOP.2010.000076. PMID 21532814